CLINICAL TRIAL: NCT01334398
Title: A Health & Wellness Intervention for Individuals With Traumatic Brain Injury
Brief Title: A Health & Wellness Intervention for Individuals With Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Craig Hospital (Other)
Responsible Party: Principal Investigator, Lisa Brenner, Director, MIRECC, VA Eastern Colorado Health Care System
Other Study IDs: 07-1146; H133A070022 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Initial Treatment Group
  Interventions: Behavioral: Health & Wellness
- Deferred Treatment Group
  Interventions: Behavioral: Health & Wellness

INTERVENTIONS:
Behavioral: Health & Wellness — The specific content of the intervention was adapted from four existing evidence-based interventions: (1) "Healthy Lifestyles for People with Disabilities," (2) Promoting Wellness for Women with MS," (3) "Living Well with Disability," and (4) "Social Skills and TBI: A Workbook for Group Treatment."

SUMMARY:
The primary goal of the proposed study is to evaluate the efficacy of a replicable community-based group intervention, designed to address both general wellness and specific TBI health-related issues. Emphasis is placed on goal setting to develop healthy habits, utilizing problem solving strategies, learning means of maintaining progress and setting new goals. Facilitators will utilize approaches aimed at maximizing participant self-efficacy, reducing barriers to health promotion, and developing personal resources. A randomized wait-list control group design will be used to evaluate the efficacy of the intervention. It is hypothesized that individuals with TBI who participate in the intervention group will report increased health promoting behaviors, health related self-efficacy, health-related quality of life, level of participation, and greater perceived wellness and satisfaction with life as compared to the control group.

DETAILED DESCRIPTION:
Health promotion in the general population and in disability groups, such as individuals with TBI, has been identified in recent decades as a specific need by the Surgeon General, the U.S. Department of Health and Human Services Healthy People 2010, the NIDRR Rehabilitation Research and Training Center (RRTC) on Health and Wellness and the Centers for Disease Control and Prevention (CDC). Additionally, decreased quality of life and increased health-related secondary conditions in TBI supports the need for health and wellness promotion. A number of health and wellness programs have been developed for specific disabled populations, with a few providing evidence for efficacy; however, no evidence based program designed to meet the unique needs of individuals with TBI has been identified. This proposal responds to the NIDRR Long Range Plan and the Healthy People 2010 call for further research in health promotion to improve quality of life, decrease disability, and eliminate disparities in health within disability populations, specifically those individuals with TBI.

The primary goal of the proposed study is to evaluate the efficacy of a replicable community-based group intervention, designed to address both general wellness and specific TBI health-related issues. Emphasis is placed on goal setting to develop healthy living habits, utilize problem solving strategies, learn means of maintaining progress and set new goals. Facilitators will utilize approaches aimed at maximizing participant self-efficacy, reducing barriers to health promotion, and developing personal resources. A randomized wait-list control group design will be used to evaluate the efficacy of the intervention.

It is hypothesized that individuals with TBI who participate in the intervention group will report increased health promoting behaviors, health related self-efficacy, health-related quality of life, level of participation, and greater perceived wellness and satisfaction with life, than the control group. Intervention group members are expected to attain individualized health and wellness goals, and maintain gains on follow-up at six months. Findings from this study will advance knowledge regarding health and wellness intervention for individuals with TBI, and may clarify areas of future research.

ELIGIBILITY:
Inclusion Criteria:

* individuals will be included in the study if they meet the following criteria:

  1. history of TBI as defined as damage to brain tissue caused by an external mechanical force as evidenced by loss of consciousness or post traumatic amnesia (PTA) due to brain trauma or by objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination.
  2. received inpatient or outpatient rehabilitation, or an evaluation related to their TBI;
  3. are classified as moderate to severe TBI based on a TBI medical/professional evaluation;
  4. are at least one year post-injury;
  5. are 18 years of age or older at the time of the study;
  6. function at Rancho Los Amigo Level of Cognitive Functioning Level of 6 or above, based on current interview with participant and family member/identified resource person
  7. have adequate receptive and expressive communication skills functional for group participation (score >5 on the Comprehension and Expression items of the Functional Independence Measure (FIM) based on current interview);
  8. have sufficient recall of day-to-day events for learning in the group setting, based on screening interview with family member or identified resource person;
  9. have the ability to participate in ongoing group sessions with no documented or reported medical or neurological conditions (e.g. upcoming hospitalizations, uncontrolled seizures), behavioral concerns (e.g. frustration tolerance, behavioral/anger control,) or other issues that preclude group participation;
  10. be English speaking in order to complete study measures (if the intervention is proven efficacious, future studies would be needed with non-English speaking participants);
  11. provide informed consent to participate.

Exclusion Criteria:

* Failure to meet inclusion criteria
* Failure to provide informed consent as evidenced by inability to respond to the above stated questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans and community members
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Health Promoting Lifestyle Profile-II | Baseline and Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, Ph.D., Principal Investigator — VA VISN 19, ECHCS; Cynthia Braden (nee Dahlberg), MA, Principal Investigator — Craig Hospital
Locations (1):
- VA ECHCS, Denver, Colorado, United States